CLINICAL TRIAL: NCT02775695
Title: Efficacy of Doxycycline on Metakaryote Cell Death in Patients With Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susan Tsai, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO28944
Record Dates: First submitted 2016-05-05; First posted 2016-05-18 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Resectable Pancreatic Cancer
Keywords: pancreatic cancer; Resectable Pancreatic Cancer; Doxycycline; Metakaryote cells; Eukaryotic cells; Cancer Stem Cells; Targeted Cancer Stem Cell Therapy; Multi-metakaryocide therapy; Doxycycline Hyclate; Tetracycline
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Doxycycline Administered to Patients (Experimental): Patients will receive oral doxycycline and trough serum concentrations for pharmacokinetic studies will be obtained.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Treatment with doxycycline hyclate will be administered as an oral agent on an outpatient basis. Patients will receive doxycycline 100 mg twice daily for a period of 8 weeks (56 days). Upon registration (baseline) and at the first, third, and fifth days of doxycycline therapy, patients will be seen to obtain trough serum concentrations for pharmacokinetic studies. Additional serum levels will be checked on days 8, 15, 22 and 29.
  Other Names: Vibramycin; Doryx

SUMMARY:
This is a window-of-opportunity study that examines the efficacy of doxycycline, and FDA-approved oral antibiotic, on metakaryotic (cancer stem cells) in resectable pancreatic cancer following eight weeks of treatment.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Pancreatic tumors have two distinct cell populations -- eukaryotic tumor cells and metakaryotic cells. The first cell type divides quickly but must stop at a certain point. Metakaryotic cells, also called cancer stem cells, divide less frequently but have an unlimited number of cell divisions. Chemotherapy works well on eukaryotic cells. Metakaryotic cells are resistant to chemotherapy and radiation, so they are more difficult to eliminate.

Massachusetts Institute of Technology basic science researchers working with the Medical College of Wisconsin pancreatic cancer group demonstrated in the laboratory that doxycycline can kill both eukaryotic and metakaryotic cells.

This study's goal is to discover if the metakaryocidal drug doxycycline kills any significant fraction of the metakaryotic cells found in treated pancreatic tumors. Targeting metakaryotic cells may decrease cancer relapse and metastases. The development of antimetakaryotics is vital for pancreatic cancer patients, who are at risk for disease recurrence and cancer-related death.

STUDY OBJECTIVES:

Primary Objectives:

To assess the efficacy of doxycycline on inducing metakaryotic cell death in primary pancreatic tumors from patients with resectable pancreatic cancer.

Secondary Objectives:

* To determine the plasma drug concentrations of the study drug at baseline and at days 1, 3, 5, 8, 15, 22, 29, and at restaging and at the time surgery.
* To assess the histopathologic treatment response of the primary tumors which have undergone neoadjuvant gemcitabine based chemoradiation and concurrent doxycycline therapy.
* To enumerate the number of observed dead/dying metakaryotes per 1 gram of resected pancreatic tissue.

STUDY PROCEDURES:

Patients will take 100 mg doxycycline twice daily for a period of eight weeks (56 days). Following standard-of-care (not study trial-related) chemotherapy, patients will receive radiation therapy. Patients will receive doxycycline beginning on the first day of radiation therapy. Following this, patients will undergo surgery four to five weeks after completion of chemoradiation. Doxycycline will be discontinued five to seven days prior to surgery.

This study involves pharmacokinetic studies, which means that patients will have blood draws several times so that serum levels may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma which may be acquired using a fine needle aspiration.
* Not received any prior therapy.
* Established resectable pancreatic cancer based on radiographic imaging.
* Patients who will receive neoadjuvant therapy (chemoradiation) are eligible.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%).
* Have no active or chronic infection with HIV, Hepatitis B or Hepatitis C
* Life expectancy of greater than six months.
* Ability to understand and the willingness to sign a written informed consent document.
* Normal organ and marrow function as defined below:

  1. leukocytes ≥3,000/microliter (mcL)
  2. absolute neutrophil count ≥1,500/mcL
  3. platelets ≥100,000/mcL
  4. total bilirubin < 2 mg/dL or has demonstrated progressive decline within two weeks of biliary decompression to allow for appropriate gemcitabine dose modification.
  5. Aspartate Aminotransferase (AST)[Serum Glutamic Oxaloacetic Transaminase (SGOT] )/ Alanine Aminotransferase (ALT) [Serum Glutamic Pyruvic Transaminase(SGPT)] ≤3 × institutional upper limit of normal
  6. Creatinine clearance ≥60 mL/min/1.73 m^2

Exclusion Criteria:

* Patients with more clinically advanced pancreatic cancer (borderline resectable, locally advanced, or metastatic).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the effects of metakaryocidal agents have the potential for teratogenic or abortifacient effects.
* Previous history of other malignancy (other than cured basal or squamous cell carcinoma of the skin or cured in-situ carcinoma of the cervix) within two years of study enrollment.
* Active or chronic HIV, hepatitis B or hepatitis C.
* Patients who are receiving other investigational drugs or enrolled in other clinical trials.
* Inability to undergo scheduled blood acquisition per protocol.
* Drug specific exclusion including history of allergic reactions to tetracyclines.
* Prior treatment with doxycycline within a seven day washout period prior to initiating treatment with alternate antimetakaryocidal medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tsai, MD, MHS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen subjects were consented to participate in the study. Three did not meet eligibility criteria during screening.
Period: Overall Study
Arm/Group | Doxycycline Administered to Patients
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Doxycycline Administered to Patients
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine the Efficacy of Doxycycline in Inducing Metakaryotic Cell Death in Primary Pancreatic Tumors as Measured by Pathologic Response
Description: The histopathologic response of the primary tumor will be assessed using the College of American Pathology criteria for residual tumor response following neoadjuvant therapy for the exocrine pancreas. Researchers will enumerate the number of observed dead/dying metakaryotes per 1 gram of resected pancreatic tissue.
Time Frame: Month 3 visit
Measure: Mean (Standard Deviation); unit: Cells/g
Arm/Group | Doxycycline Administered to Patients
Number analyzed (Participants) | 12
Cells/g | 8.9 (7.25)

ADVERSE EVENTS:
Time Frame: Each participant was assessed from adverse events up to a maximum of 1 year.
Arm/Group | Doxycycline Administered to Patients
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline Administered to Patients (N=12)
Anaphylaxis (Immune system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - other, specify (Gastrointestinal disorders) | 2 (2)
Ascities (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline Administered to Patients (N=12)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Ascities (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomitiing (Gastrointestinal disorders) | 1 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (18)
Neutrophil count decreased (Investigations) | 6 (7)
Platelet count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT02775695/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT02775695/ICF_001.pdf